CLINICAL TRIAL: NCT00707551
Title: A Phase I, Single-centre, Randomised, Open, Three-way Crossover Study to Evaluate the Effect of Ketoconazole and Verapamil, Respectively, on the Pharmacokinetics of AZD1305 After Repeated Oral Adm of Ketoconazole and Verapamil and Single Oral Dosing of AZD1305 to Young Healthy Male Volunteers
Brief Title: An Interaction Study of Ketoconazole/Verapamil Versus AZD1305
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Helen Lunde, MD, Medical Science Director, Emerging Arrhythmia and Lipids, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D3190C00009; 2008-000578-18 (EudraCT No)
Record Dates: First submitted 2008-06-27; First posted 2008-07-01 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: AZD1305; Verapamil; Ketoconazole; pharmacokinetics
MeSH Terms: interventions — Ketoconazole; Verapamil; tert-butyl (2-(7-(2-(4-cyano-2-fluorophenoxy)ethyl)-9-oxa-3,7-diazabicyclo(3.3.1)non3-yl)ethyl)carbamate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Ketoconazole tablet + AZD1305 Extended Release tablet
  Interventions: Drug: Ketoconazole; Drug: AZD1305
- 2 (Experimental): Verapamil Extended Release tablet + AZD1305 Extended Release tablet
  Interventions: Drug: Verapamil; Drug: AZD1305
- 3 (Experimental): AZD1305 Extended Release tablet
  Interventions: Drug: AZD1305

INTERVENTIONS:
Drug: Ketoconazole — Tablet, administered as repeated doses.
  Other Names: Fungoral
  Arms: 1
Drug: Verapamil — Extended Release tablet, administered as repeated doses.
  Other Names: Isoptin Retard
  Arms: 2
Drug: AZD1305 — Extended Release tablet, administered as a single dose.

SUMMARY:
The purpose is to study whether ketoconazole or verapamil have an effect on how AZD1305 is handled by the body, i.e the absorption, distribution, metabolism and excretion, when administered in combination with AZD1305.

ELIGIBILITY:
Inclusion Criteria:

* A body mass index (BMI=weight/height2) of 19 to 30 kg/m2

Exclusion Criteria:

* Potassium outside normal reference values
* ECG findings outside normal range

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic variables | During all dosing visits

SECONDARY OUTCOMES:
Adverse events, vital signs, ECG, laboratory variables and physical examination | During the study

CONTACTS AND LOCATIONS:
Overall Officials: Helen Lunde, MD, Study Director — AstraZeneca R&D, Mölndal, Sweden; Dago Mazur, MD, PhD, Principal Investigator — PAREXEL International GmbH, Berlin, Germany
Locations (1):
- Research Site, Berlin, Germany